CLINICAL TRIAL: NCT06879236
Title: Secondary and Tertiary Digital Prevention of Non-alcoholic and Dysmetabolic Liver Disease
Acronym: CALIBRE
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 6618
Record Dates: First submitted 2024-09-26; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: NASH; NAFLD
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The prevalence of Metabolic dysfunction-associated steatotic liver disease (MASLD) and its severe form, Metabolic dysfunction-associated steatohepatitis (MASH), is high and they are increasingly becoming major causes of cirrhosis, hepatocellular carcinoma (HCC), and the need for liver transplantation. Due to the lack of noticeable symptoms during the early stages, the detection of MASLD is often delayed until the disease has advanced.

Currently, the treatment options MASLD are limited to lifestyle interventions such as dietary changes and physical activity. Despite the increasing prevalence of MASLD, there are no drugs available on the market specifically for this condition.

The goal is to made new model care which integrates the standard clinical procedures with a digital approach, namely a mobile application for patients and a clinical dashboard for healthcare professionals (HCPs), integrated with simple clinical data (anthropometric, laboratory and imaging data).

This study wants to test the feasibility of integrating a digital intervention to improve the patient engagement and linkage to care in order to identify the advanced MASLD at earliest stage (secondary prevention) and mitigate the impact of ongoing advanced liver disease helping patients to manage the long-term effect of disease.

To achieve this goal the study will leverage on a mobile app named OpenTele in order to test the adherence to lifestyle changes in patient with MASLD and on the connected clinical dashboard.

The app aims at integrating the standard clinical practice with digital technologies able to guide and support patients in order to seamlessly integrate secondary prevention strategies in their everyday life with 2 main aims:

* to implement a strategy for delay progression of liver disease;
* to reduce the effect of cirrhosis (tertiary prevention).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with MASLD and LSM>= 10 kPa
* Age >= 18 years old
* Sufficient digital literacy or supported from a caregiver with sufficient digital literacy
* Smartphone (Android or iOS) able to download and run the App
* Able to understand and communicate in Italian
* Able to sign the informed consent

Exclusion Criteria:

* Major psychiatric disorder
* Not able to use digital technologies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: subjects with type 2 diabetes and/or metabolic syndrome and/or dyslipidemia and/or obesity (BMI>30 Kg/m2) and/or familiar history for cirrhosis or liver cancer in the absence of known risk factors
Sampling Method: Probability Sample
Enrollment: 252 (Estimated)
Dates: Start 2025-01-16 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
App Adherence (>80% over 4 weeks) | 4 weeks
  Assessed via smartphone (number of app access)

SECONDARY OUTCOMES:
Weight reduction assessment | 12 month
  Number of subjects with a 12-month reduction between 7-10% of weight compared to baseline
Change in liver and spleen stiffness | Baseline, after 4 weeks and 12 month
  Assessed by transient elastography
Change in Patient Reported Outcome questionnaire | 12 weeks
  Evaluation of overall physical well-being through the administration of questionnaires
Changes in measure energy expenditure | 12 month
  Cycle ergometer
Microbiome signature | 12 month
  Analysis of microbiome signature from feces
Clinical events | 12 month
  Record of number of hospitalization, decompensation, variceal bleeding, encephalopathy, ascites, liver cancer, liver transplantation, death

CONTACTS AND LOCATIONS:
Overall Officials: Luca Miele, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, UOC Medicina Trapianti Fegato and UOC CEMAD, Rome, Lazio, Italy